CLINICAL TRIAL: NCT04357483
Title: Randomized Controlled Study to Evaluate the Effect of Thrombin-containing Collagen-based Hemostatic Matrix on Prevention of Pancreatic Fistula After Pancreatecomy
Brief Title: Effect of Thrombin-containing Collagen-based Hemostatic Matrix
Acronym: TCM
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Song Cheol Kim, Director, Asan Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Collastat 2020
Record Dates: First submitted 2020-04-20; First posted 2020-04-22 (Actual); Last update posted 2020-04-28 (Actual); Status verified 2020-04

CONDITIONS: Pancreatic Tumor
Keywords: Postoperative pancreatic fistula; Pancreatectomy
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Collagen

STUDY DESIGN:
Intervention Model Description: Arm1 (intervention) : flowable thrombin containing collagen hemostat matrix Arm2 (Control) : thrombin coated L-dopa contained collagen patch
Who Masked: Participant
Masking Description: Single Blind
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Collastat (Experimental): Patients who were applied flowable thrombin containing collagen hemostat matrix after pancreatectomy
  Interventions: Drug: flowable thrombin containing collagen hemostat matrix
- Collaseal (Active Comparator): Patients who were applied thrombin coated L-dopa contained collagen patch after pancreatectomy
  Interventions: Drug: thrombin coated L-dopa contained collagen patch

INTERVENTIONS:
Drug: flowable thrombin containing collagen hemostat matrix — A 5 ml flowable hemostat matrix (CollaStat®) was applied to the stump or anastomosis site after pancreatectomy.
  Other Names: CollaStat®
  Arms: Collastat
Drug: thrombin coated L-dopa contained collagen patch — A 5x2.5cm sized thrombin coated L-dopa contained collagen patch (CollaSeal®) was applied to the stump or anastomosis site after pancreatectomy.
  Other Names: CollaSeal®
  Arms: Collaseal

SUMMARY:
Under the hypothesis that collagen-based hemostatic agents improve the suppression of leakage of hemostatic pancreatic fluid at the surgical site during surgery, thrombin-containing collagen-based hemostatic agents are applied in surgery in patients with pancreatectomy. The investigators intend to evaluate the effectiveness of collagen-based hemostatic agents containing thrombin through clinical evaluation of hemostatic effect and anti-leakage effect of pancreatic fluid.

This clinical study is a study for comparative evaluation of hemostasis and anti-leakage effect of bile or pancreatic fluid when applied after pancreatic resection of a collagen-based hemostatic agent containing thrombin. It is prospective, single center, randomized, and non-inferiority test. Participants are patients who are diagnosed with pancreatic disease and other diseases, and plan to undergo pancreatectomy. Through the randomization, in the case of the intervention group, after the pancreatectomy, the Collastat (CollaStat®, Dalim Tissen. Co., Ltd., Korea) is applied to the cut surface, and in the case of the control group, Collaseal (CollaSeal®, Dalim Tissen. Co., Ltd., Korea) is applied. In this study, 30 participants were required for each intervention group and control group.

After surgery, the participants is hospitalized for 7 days and undergoes follow-up observation. Pancreatic leakage is measured through the drainage tube before discharge and evaluated as biochemical leakage (BL), B, or C according to the definition of International Study Group for Pancreatic Fistula (ISGPS).

The primary endpoint of this study was the prevention rate of leakage. The postoperative pancreatic fistula (POPF) was defined according to the definition of ISGPS. Secondary end point was assessed as the difference between groups of total number of collagen hemostatic agents used, hospital length of stay and number of patient who received RBC transfusion. Safety was assessed based on the incidence of adverse events occurred.

DETAILED DESCRIPTION:
1. Synopsis

   * Title: Randomized controlled Study to evaluate the Effect of Thrombin-containing Collagen-based Hemostatic Matrix on Prevention of Pancreatic fistula after Pancreatectomy
   * Study center: Single center from Korea
   * Study type: Single center prospective randomized controlled study
   * Planned study dates: February 2018 to September 2020
2. Objectives

   ■ The aim of this study was to evaluate the safety and efficacy of flowable thrombin containing collagen hemostat matrix (T-C matrix) over the thrombin coated L-dopa contained collagen patch (T-CD patch) on clinical outcomes including PPH and POPF as a randomized controlled clinical trial.
3. Background

   * Hemostasis is the most basic and important procedure as a treatment for bleeding that inevitably follows most surgical procedures. Recently, with the development of pancreatic surgery and postoperative management, the mortality rate associated with surgery has decreased significantly, but the rate of complications due to massive bleeding or leakage of pancreatic fluid during surgery has not changed significantly. In hepatobiliary and pancreas (HBP) surgery, post-pancreatectomy hemorrhage (PPH) and postoperative pancreatic fistula (POPF) are both the main source of major morbidity and mortality.
   * Collagen is a natural substrate for various kinds of animal cells, and contains a relatively large amount compared to other proteins in animal tissues, and can be easily extracted and purified from animal tissues. Collagen not only has low antigenicity, but also has excellent hemostatic effect and cell attachment ability, so it is often used as a major component of hemostatic agents and artificial tissue substitutes. In addition, collagen provides an environment in which fibroblasts can be produced and induces wound healing by inactivating elastase and matrix metalloproteases (MMPs).
   * The investigators developed a novel flowable thrombin containing collagen hemostat matrix (T-C matrix) having flowable paste-like form. The T-C matrix consists of two connectable syringes, one of which contains collagen granules and thrombin, and the other contains calcium chloride (CaCl2) solution. Due to the flowable characteristic of the resultant matrix, T-C matrix can be easily applicable to irregular surface such as surgical site where anastomotic leakage is a concern. Currently, thrombin /coated L-3,4-dihydroxyphenylalanine (L-dopa DOPA) contained collagen patch (T-CD patch) are using on prevention of leakage and bleeding in pancreatic surgery. Although L-DOPA is known to contribute to adhesiveness which facilitates application of T-CD patch on wound sites, there are some controversial studies that L-DOPA have cytotoxicity and may induce inflammatory reaction with a high dose.
4. Methodology

   * The clinical study was designed to evaluate the effect of T-C matrix on the prevention of leakage in a pancreatectomy. The expected number of participants is 60.
   * This clinical study is a randomized prospective comparative study of the outcome according to the hemostat materials as a non-inferiority test, and the research hypothesis is as follows.

     √ Null Hypothesis: There is no difference in the incidence of POPF between patients who were applied TC matrix (CollaStat®, Dalim Tissen. Co., Ltd., Korea) and T-CD patch (CollaSeal®, Dalim Tissen Co. Ltd., Korea) after pancreatectomy.
   * In the case of evaluating the incidence of POPF after pancreatectomy, the results of previous studies of the 'leakage' ratio showed a leak prevention effect (θA) = 88% of the existing treatment method of CollaSeal® analog (Montorsi M et al. 2012). The new treatment effect (θT) is intended to demonstrate non-inferiority that does not exceed the non-inferiority limit (δ) compared to the existing treatment effect (θA). The non-inferiority limit (δ) was calculated by more than 75% of the existing treatment effect. The non-inferiority limit was calculated to be 0.22 based on the case where more than 75% of the 88% of the existing treatment method is confirmed, that is, the treatment success rate is more than 66%. It was decided that CollaStat® was non-inferior to CollaSeal® when the lower limit of the 95% CI for the difference between the two groups was greater than -0.22. If the allocation ratio between the two groups is 1: 1 and the first-class error α = 5% and the second-class error β = 20%, considering the dropout rate of 10%, 30 study groups and control groups each need 30 subjects.
   * The random assignment of this study is assigned according to the order of assignment in the planning stage of the study as a block randomization scheme with appropriate block size set.

ELIGIBILITY:
Inclusion Criteria:

* Age: 20-80 years at the day of enrollment
* Performance: ECOG 0-2
* Patients who was scheduled for pancreatectomy due to benign or malignant tumor
* No distant metastasis
* Bone marrow function: WBC at least 3,000 / mm3, Platelet count at least 100,000 / mm3
* Liver function: AST / ALT less than 3 times upper limit of normal
* Kidney function: Creatinine no greater than 1.5 times upper limit of normal.
* Patients who consented to and signed the consent

Exclusion Criteria:

* Those with active or uncontrolled infections
* Those with severe psychiatric / neurological disorders
* Alcohol or other drug addicts
* Patients included in other clinical studies that may affect this study
* Patients who cannot follow the directions of the researcher
* Those with uncontrolled heart disease
* Patients with moderate or severe comorbidities who are thought to have an impact on quality of life or nutritional status (cirrhosis, chronic kidney failure, heart failure, etc.)
* Pelvic tumor, benign tumor, malignant tumor in other organs
* pregnant or planning on becoming pregnant during the follow-up period
* undergoing lymphatic or coagulation disease
* known sensitivity or allergy to bovine and/or porcine substance(s)

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2018-02-01 (Actual); Primary Completion 2020-07-31 (Estimated); Study Completion 2020-09-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of POPF | Three months
  Pancreatic leakage is measured through the drainage tube before discharge and evaluated as biochemical leakage (BL), B, or C according to the definition of International Study Group for Pancreatic Fistula (ISGPS).

SECONDARY OUTCOMES:
hospital length of stay | Three months
  The length of hospital stay after surgery is observed.
number of patient who received RBC transfusion | One months
  The amount of blood transfusion performed during surgery should be described.
Postoperative complication | Three months
  According to the Clavien-Dindo classification, the grade of complication including readmission should be described.

CONTACTS AND LOCATIONS:
Overall Officials: Song Cheol Kim, MD, PhD, Study Chair — Asan Medical Center
Locations (1):
- Asan medical center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Schwartz M, Madariaga J, Hirose R, Shaver TR, Sher L, Chari R, Colonna JO 2nd, Heaton N, Mirza D, Adams R, Rees M, Lloyd D. Comparison of a new fibrin sealant with standard topical hemostatic agents. Arch Surg. 2004 Nov;139(11):1148-54. doi: 10.1001/archsurg.139.11.1148. PMID 15545559
- [Background] Zegers M, de Bruijne MC, de Keizer B, Merten H, Groenewegen PP, van der Wal G, Wagner C. The incidence, root-causes, and outcomes of adverse events in surgical units: implication for potential prevention strategies. Patient Saf Surg. 2011 May 20;5:13. doi: 10.1186/1754-9493-5-13. PMID 21599915
- [Background] Chiara O, Cimbanassi S, Bellanova G, Chiarugi M, Mingoli A, Olivero G, Ribaldi S, Tugnoli G, Basilico S, Bindi F, Briani L, Renzi F, Chirletti P, Di Grezia G, Martino A, Marzaioli R, Noschese G, Portolani N, Ruscelli P, Zago M, Sgardello S, Stagnitti F, Miniello S. A systematic review on the use of topical hemostats in trauma and emergency surgery. BMC Surg. 2018 Aug 29;18(1):68. doi: 10.1186/s12893-018-0398-z. PMID 30157821
- [Background] Suzuki Y, Kuroda Y, Morita A, Fujino Y, Tanioka Y, Kawamura T, Saitoh Y. Fibrin glue sealing for the prevention of pancreatic fistulas following distal pancreatectomy. Arch Surg. 1995 Sep;130(9):952-5. doi: 10.1001/archsurg.1995.01430090038015. PMID 7661678
- [Background] Wilson C, Robinson S, French J, White S. Strategies to reduce pancreatic stump complications after open or laparoscopic distal pancreatectomy. Surg Laparosc Endosc Percutan Tech. 2014 Apr;24(2):109-17. doi: 10.1097/SLE.0b013e3182a2f07a. PMID 24686344
- [Background] Rickenbacher A, Breitenstein S, Lesurtel M, Frilling A. Efficacy of TachoSil a fibrin-based haemostat in different fields of surgery--a systematic review. Expert Opin Biol Ther. 2009 Jul;9(7):897-907. doi: 10.1517/14712590903029172. PMID 19527109
- [Background] Hiura Y, Takiguchi S, Yamamoto K, Kurokawa Y, Yamasaki M, Nakajima K, Miyata H, Fujiwara Y, Mori M, Doki Y. Use of fibrin glue sealant with polyglycolic acid sheets to prevent pancreatic fistula formation after laparoscopic-assisted gastrectomy. Surg Today. 2013 May;43(5):527-33. doi: 10.1007/s00595-012-0253-2. Epub 2012 Jul 14. PMID 22797962